CLINICAL TRIAL: NCT01568853
Title: The Complement C3 Depletion in Patients With Severe Abdominal Sepsis: Risk Prediction and the Association With Down-regulated Adaptive Immunity
Brief Title: A Prospective Study of The Complement Depletion in Patients With Severe Abdominal Sepsis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Jianan Ren, Clinical professor, Principal investigator, Jinling Hospital, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: BK2010-017-1
Record Dates: First submitted 2012-03-29; First posted 2012-04-02 (Estimated); Last update posted 2012-04-06 (Estimated); Status verified 2012-04

CONDITIONS: Severe Sepsis; Pancreatitis; Abdominal Abscess; Appendicitis; Digestive System Fistula
MeSH Terms: conditions — Sepsis; Pancreatitis; Abdominal Abscess; Appendicitis; Digestive System Fistula | interventions — Norepinephrine; Open Abdomen Techniques; Enteral Nutrition; Parenteral Nutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Norepinephrine — Intravenously, 10 ug/min, 24 hours
Procedure: Open abdomen — IAH >=20 mmHg, and ACS emerged, such as low urine and decreased FiO2 quickly.
Other: enteral nutrition — 500-1500 kcal/day; Nasogastric tube feeding;
  Other Names: Peptison (SP; Nutricia, Shanghai, China)
Other: parenteral nutrition — 3000 mL parenteral nutrition fluid, intravenously.
  Other Names: Made by our hospital.

SUMMARY:
The role of complement system in bridging innate and adaptive immunity has been confirmed in various invasive pathogens. The aim of this study is to investigate the alteration of complement C3 in patients with severe abdominal sepsis and evaluate the role of complement C3 depletion in prognosis of such patients. The relationship between complement C3 depletion and adaptive immunity is studied meanwhile.

DETAILED DESCRIPTION:
Severe abdominal sepsis remains a significant cause of death in patients undergoing intra-abdominal infection, in despite of recent declines in overall mortality. There is a abundant evidence to suggest complement activation during sepsis. While there is great interest in complement by-products in human sepsis, few studies focus on the persistent consumption of complement components and its role in prognosis of sepsis. Complement C3 is indispensable community pathway for complement activation. In a way, the alteration of C3 levels can affect the whole status of complement biological functions.

In clinical practice, the severe abdominal sepsis would develop compromised immune function if the intra-abdominal infection is not well controlled. The down-regulated T- and B-cell immune responses to sepsis are correlated to the decreased immune defense. To our knowledge, there are few human data that have investigated the relationship between complement depletion and adaptive immunity in severe abdominal sepsis. The investigators hypothesize that the complement C3 depletion during sepsis has a stronger association with the down-regulated adaptive immunity and can be regarded as a essential risk factor to predict the prognosis of such critical illness.

The purpose of this prospective study is two-fold. First, the investigators observe, in a cohort of patients with severe abdominal sepsis, the levels of complement components and percentages of T cell subsets after admission to evaluate the relationship between complement system and adaptive immunity. Second, the investigators also evaluate the application of the C3 related-indexes (C3, C3a, Factor H, DAF, etc.) to patients undergoing severe abdominal sepsis and to develop an alternative model to predict its prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of severe abdominal sepsis

Exclusion Criteria:

* Age < 18 or > 60 years
* Pregnancy
* Leucopenia from radiochemical therapy due to malignant tumor
* Any primary diagnosis other than sepsis
* Confirmed immunodeficiency
* Requirement for blood transfusion, plasmapheresis, or immediate surgery

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2011-11; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
All cause mortality | within the first 28 days after admission to our hosptial
  Patients died within the first three days of admission would be excluded from this study.

SECONDARY OUTCOMES:
Postoperative complications | within the first 28 days after admission to our hosptial
  wound complications; pulmonary infection; incisional hernia, and bleeding.

CONTACTS AND LOCATIONS:
Overall Officials: Jianan Ren, M.D., Principal Investigator — Department of Surgery, Jinling Hospital, China
Locations (1):
- Department of Surgery, Jinling Hospital, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Ren J, Zhao Y, Yuan Y, Han G, Li W, Huang Q, Tong Z, Li J. Complement depletion deteriorates clinical outcomes of severe abdominal sepsis: a conspirator of infection and coagulopathy in crime? PLoS One. 2012;7(10):e47095. doi: 10.1371/journal.pone.0047095. Epub 2012 Oct 16. PMID 23091606